CLINICAL TRIAL: NCT03465878
Title: A Study to Evaluate the Pharmacokinetics and Glucodynamics of LY900014 Compared to Humalog in Children, Adolescents, and Adults With Type 1 Diabetes Mellitus
Brief Title: A Study of LY900014 in Participants With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16695; I8B-MC-ITSA (Other: Eli Lilly and Company); 2017-003220-78 (EudraCT Number)
Record Dates: First submitted 2018-03-09; First posted 2018-03-14 (Actual); Results first posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2019-12

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY900014-Part A (Experimental): Participants received single 0.2 U/kg of body weight subcutaneous (SC) bolus injection of 100 U/mL LY900014.
  Interventions: Drug: LY900014
- Humalog (Insulin Lispro)-Part A (Active Comparator): Participants received single 0.2 U/kg of body weight SC bolus injection of 100 U/mL of Humalog.
  Interventions: Drug: Insulin Lispro
- LY900014-Part B (Experimental): Participants received single 0.2 U/kg of body weight SC bolus infusion of 100 U/mL LY900014 delivered using the continuous subcutaneous insulin infusion (CSII) pump.
  Interventions: Drug: LY900014
- Humalog (Insulin Lispro)-Part B (Active Comparator): Participants received single 0.2 U/kg of body weight SC bolus infusion of 100 U/mL Humalog delivered using the CSII pump.
  Interventions: Drug: Insulin Lispro

INTERVENTIONS:
Drug: LY900014 — Administered via SC injection
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014-Part A; LY900014-Part B
Drug: Insulin Lispro — Administered via SC injection
  Other Names: Humalog; LY275585
  Arms: Humalog (Insulin Lispro)-Part A; Humalog (Insulin Lispro)-Part B

SUMMARY:
The purpose of this study is to compare LY900014 with insulin lispro (Humalog) in participants with type 1 diabetes mellitus.

There are 2 parts to this study. Part A is investigating how the body processes LY900014 and the effect of LY900014 on blood sugar levels compared to insulin lispro (Humalog) when study treatment is given by subcutaneous injection. Part B of the study is investigating how the body processes LY900014 and the effect of LY900014 on blood sugar levels compared to insulin lispro (Humalog) when study treatment is given by continuous subcutaneous insulin infusion (CSII) pump.

Screening is required within 28 days prior to the start of the study. For each participant, the study will last about 40 days in each part.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female participants aged 6-64 with Type 1 Diabetes Mellitus (T1DM) for at least 1 year
* Have a glycated hemoglobin (HbA1c) less than (<)10.0 percent (%)

Exclusion Criteria:

* Receiving any oral or injectable medication intended for the treatment of diabetes mellitus other than insulins in the 12 months prior to screening
* More than one episode of severe hypoglycaemia in the last 6 months
* Presence of clinically significant hematologic, oncologic, renal, cardiac, hepatic, or gastrointestinal disease, proliferative retinopathy, uncontrolled celiac disease, uncontrolled hyperthyroidism or hypothyroidism, or adrenal insufficiency
* Have obvious clinical signs or symptoms of liver disease
* Have a history of renal impairment

Ages: 6 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- LMC Endocrinology Centres Ltd., Toronto, Ontario, Canada
- Kinderkrankenhaus auf der Bult, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY900014 in Participants With Type 1 Diabetes Mellitus — https://www.lillytrialguide.com/en-US/studies/type-1-diabetes/ITSA#?postal=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (pts) who completed Part A but discontinued before the beginning of Part B were replaced by newly enrolled participants in Part B.
Pre-assignment Details: Two period crossover study, with a minimum of 22 days washout period between each period.
Groups:
- Sequence 1-Part A: Participants received either single 0.2 units per kilogram (U/kg) of body weight subcutaneous (SC) bolus injection of 100 units per milliliter (U/mL) LY900014 or Humalog.
  Period 1: LY900014 Period 2: Humalog
- Sequence 2-Part A: Participants received either single 0.2 U/kg of body weight subcutaneous (SC) bolus injection of 100 U/mL LY900014 or Humalog.
  Period 1: Humalog Period 2: LY900014
- Sequence 1-Part B: Participants received either single 0.2 U/kg of body weight subcutaneous (SC) bolus infusion of 100 U/mL LY900014 or Humalog delivered using the continuous subcutaneous insulin infusion (CSII) pump.
  Period 1: LY900014 Period 2: Humalog
- Sequence 2-Part B: Participants received either single 0.2 U/kg of body weight subcutaneous (SC) bolus infusion of 100 U/mL LY900014 or Humalog with delivered using the CSII pump.
  Period 1: Humalog Period 2: LY900014
Period: Period 1-Part A First Intervention Day 1
Arm/Group | Sequence 1-Part A | Sequence 2-Part A | Sequence 1-Part B | Sequence 2-Part B
Started | 21 | 21 | 0 | 0
Received at Least 1 Dose of Study Drug | 21 | 21 | 0 | 0
Children (2-11 Years) | 7 | 6 | 0 | 0
Adolescents (12-17 Years) | 7 | 7 | 0 | 0
Adults (18-64 Years) | 7 | 8 | 0 | 0
Completed | 21 | 20 | 0 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Period2-Part A Second Intervention Day 1
Arm/Group | Sequence 1-Part A | Sequence 2-Part A | Sequence 1-Part B | Sequence 2-Part B
Started | 21 | 20 | 0 | 0
Children (2-11 Years) | 7 | 6 | 0 | 0
Adolescents (12-17 Years) | 7 | 7 | 0 | 0
Adults (18-64 Years) | 7 | 7 | 0 | 0
Completed | 21 | 20 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Period 1-Part B First Intervention Day 1
Arm/Group | Sequence 1-Part A | Sequence 2-Part A | Sequence 1-Part B | Sequence 2-Part B
Started | 0 (This period is for Part B group.) | 0 (This period is for Part B group.) | 20 (25 pts from Part A were re-randomized to Part B, 14 new pts were randomized in Part B.) | 19 (25 pts from Part A were re-randomized to Part B, 14 new pts were randomized in Part B.)
Received at Least 1 Dose of Study Drug | 0 | 0 | 20 | 17
Children (2-11 Years) | 0 | 0 | 6 | 6
Adolescents (12-17 Years) | 0 | 0 | 7 | 6
Adults (18-64 Years) | 0 | 0 | 7 | 5
Completed | 0 | 0 | 20 | 17
Not Completed | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1
Period: Period2-Part B Second Intervention Day 1
Arm/Group | Sequence 1-Part A | Sequence 2-Part A | Sequence 1-Part B | Sequence 2-Part B
Started | 0 | 0 | 20 | 17
Children (2-11 Years) | 0 | 0 | 6 | 6
Adolescents (12-17 Years) | 0 | 0 | 7 | 6
Adults (18-64 Years) | 0 | 0 | 7 | 5
Completed | 0 | 0 | 20 | 17
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All newly randomized participants of Part A and Part B.
Groups:
- Part A: Participants received single 0.2 U/kg of body weight SC bolus injection of 100 U/mL LY900014 or Humalog.
- Part B: Participants received single 0.2 U/kg of body weight subcutaneous (SC) bolus infusion of either 100 U/mL LY900014 or Humalog delivered using the CSII pump.
- Total: Total of all reporting groups
Arm/Group | Part A | Part B | Total
Number analyzed (Participants) | 42 | 14 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.5 (15.1) | 23.2 (11.1) | 21.2 (14.2)
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 Years) | 13 | 3 | 16
  Adolescents (12-17 years) | 14 | 2 | 16
  Adults (18-64 years) | 15 | 9 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 8 | 28
  Male | 22 | 6 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 40 | 14 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 37 | 11 | 48
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 28 | 10 | 38
  Germany | 14 | 4 | 18

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Insulin Lispro Area Under the Concentration Curve (AUC) Following Each Treatment Arm for Each Study Part
Description: Pharmacokinetics (PK): Insulin Lispro Area Under the Concentration Curve (AUC(0 -7h)) following Each Treatment Arm for Each Study Part.
Time Frame: Predose, 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 60, 70, 90, 120, 150, 180, 240, 300, 360, and 420 minutes postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picomoles*hour/Liter (pmol*h/L)
Groups:
- Children-LY900014-Part A: Participants received single 0.2 U/kg of body weight subcutaneous (SC) bolus injection of 100 U/mL LY900014.
- Children-Humalog-Part A; Adolescents-Humalog-Part A; Adults-Humalog-Part A: Participants received single 0.2 U/kg of body weight SC bolus injection of 100 U/mL Humalog.
- Adolescents-LY900014-Part A: Participants received single 0.2 U/kg of body weight SC bolus injection of 100 U/mL LY900014.
- Adults-LY900014-Part A: Participants received single 0.2 U/kg of body weight SC bolus injection of 100U/mL LY900014.
- Children-LY900014-Part B; Adolescents-LY900014-Part B; Adults-LY900014-Part B: Participants received single 0.2 U/kg of body weight SC bolus infusion of 100 U/mL LY900014 delivered using the CSII pump.
- Children-Humalog-Part B; Adolescents-Humalog-Part B; Adults-Humalog-Part B: Participants received single 0.2 U/kg of body weight SC bolus infusion of 100 U/mL Humalog delivered using the CSII pump.
Arm/Group | Children-LY900014-Part A | Children-Humalog-Part A | Adolescents-LY900014-Part A | Adolescents-Humalog-Part A | Adults-LY900014-Part A | Adults-Humalog-Part A | Children-LY900014-Part B | Children-Humalog-Part B | Adolescents-LY900014-Part B | Adolescents-Humalog-Part B | Adults-LY900014-Part B | Adults-Humalog-Part B
Number analyzed (Participants) | 13 | 13 | 14 | 14 | 14 | 14 | 11 | 11 | 13 | 13 | 12 | 12
Picomoles*hour/Liter (pmol*h/L) | 755 (15) | 754 (17) | 962 (17) | 908 (21) | 987 (20) | 975 (21) | 743 (17) | 714 (17) | 842 (20) | 866 (16) | 1100 (35) | 1070 (35)
Statistical Analysis 1: Comparison: Children-LY900014-Part A vs Children-Humalog-Part A; Test type: Superiority; p = 0.9813, Mixed Models Analysis; Ratio of geometric least squares means = 0.999, 95% CI 2-sided [0.918 to 1.09]
Statistical Analysis 2: Comparison: Adolescents-LY900014-Part A vs Adolescents-Humalog-Part A; Test type: Superiority; p = 0.1638, Mixed Models Analysis; Ratio of geometric least squares means = 1.06, 95% CI 2-sided [0.976 to 1.15]
Statistical Analysis 3: Comparison: Adults-LY900014-Part A vs Adults-Humalog-Part A; Test type: Superiority; p = 0.7623, Mixed Models Analysis; Ratio of geometric least squares means = 1.01, 95% CI 2-sided [0.933 to 1.10]
Statistical Analysis 4: Comparison: Children-LY900014-Part B vs Children-Humalog-Part B; Test type: Superiority; p = 0.2952, Mixed Models Analysis; Ratio of geometric least squares means = 1.04, 95% CI 2-sided [0.962 to 1.13]
Statistical Analysis 5: Comparison: Adolescents-LY900014-Part B vs Adolescents-Humalog-Part B; Test type: Superiority; p = 0.4052, Mixed Models Analysis; Ratio of geometric least squares means = 0.970, 95% CI 2-sided [0.901 to 1.04]
Statistical Analysis 6: Comparison: Adults-LY900014-Part B vs Adults-Humalog-Part B; Test type: Superiority; p = 0.5314, Mixed Models Analysis; Ratio of geometric least squares means = 1.02, 95% CI 2-sided [0.948 to 1.11]

2. Secondary Outcome: Glucodynamics (GD): Area Under the Baseline Subtracted Glucose Concentration Versus Time Curve Following Each Treatment Arm for Each Study Part
Description: Glucodynamics (GD): Area Under the Baseline Subtracted Glucose Concentration Versus Time Curve (BG∆AUC(0-5h)) Following Each Treatment Arm for Each Study Part.
Time Frame: -30, -15, 0 (predose), 10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 110, 120, 135, 150, 165, 180, 195, 210, 225, 240 and 300 minutes postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable Glucodynamics data.
Measure: Mean (Standard Deviation); unit: milligrams*hour per deciliter (mg*h/dL)
Arm/Group | Children-LY900014-Part A | Children-Humalog-Part A | Adolescents-LY900014-Part A | Adolescents-Humalog-Part A | Adults-LY900014-Part A | Adults-Humalog-Part A | Children-LY900014-Part B | Children-Humalog-Part B | Adolescents-LY900014-Part B | Adolescents-Humalog-Part B | Adults-LY900014-Part B | Adults-Humalog-Part B
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 14 | 14 | 10 | 10 | 13 | 13 | 12 | 12
milligrams*hour per deciliter (mg*h/dL) | 384 (335) | 492 (270) | 577 (247) | 651 (238) | 372 (179) | 351 (240) | 602 (221) | 582 (254) | 614 (160) | 614 (163) | 343 (194) | 401 (235)

ADVERSE EVENTS:
Time Frame: From Baseline to Study Completion (Up to 20 Months)
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Children-LY900014-Part A | Children-Humalog-Part A | Adolescents-LY900014-Part A | Adolescents-Humalog-Part A | Adults-LY900014-Part A | Adults-Humalog-Part A | Children-LY900014-Part B | Children-Humalog-Part B | Adolescents-LY900014-Part B | Adolescents-Humalog-Part B | Adults-LY900014-Part B | Adults-Humalog-Part B
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/14 | 0/14 | 0/14 | 0/15 | 0/12 | 0/12 | 0/13 | 0/13 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 1/14 | 0/14 | 0/14 | 0/15 | 0/12 | 0/12 | 0/13 | 0/13 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 4/13 | 4/13 | 6/14 | 3/14 | 2/14 | 2/15 | 6/12 | 4/12 | 3/13 | 1/13 | 3/12 | 2/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Children-LY900014-Part A (N=13) | Children-Humalog-Part A (N=13) | Adolescents-LY900014-Part A (N=14) | Adolescents-Humalog-Part A (N=14) | Adults-LY900014-Part A (N=14) | Adults-Humalog-Part A (N=15) | Children-LY900014-Part B (N=12) | Children-Humalog-Part B (N=12) | Adolescents-LY900014-Part B (N=13) | Adolescents-Humalog-Part B (N=13) | Adults-LY900014-Part B (N=12) | Adults-Humalog-Part B (N=12)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Children-LY900014-Part A (N=13) | Children-Humalog-Part A (N=13) | Adolescents-LY900014-Part A (N=14) | Adolescents-Humalog-Part A (N=14) | Adults-LY900014-Part A (N=14) | Adults-Humalog-Part A (N=15) | Children-LY900014-Part B (N=12) | Children-Humalog-Part B (N=12) | Adolescents-LY900014-Part B (N=13) | Adolescents-Humalog-Part B (N=13) | Adults-LY900014-Part B (N=12) | Adults-Humalog-Part B (N=12)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acne pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/78/NCT03465878/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT03465878/SAP_001.pdf